CLINICAL TRIAL: NCT04896346
Title: Scarring in Stratagraft-treated vs. Autograft-treated Burn Wounds: a Clinical and Histological Investigation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00002861
Record Dates: First submitted 2021-03-09; First posted 2021-05-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Burn Scar; Scar
Keywords: stratagraft
MeSH Terms: conditions — Cicatrix | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One 3-millimeter punch biopsy will be obtained from each subjects Stratagraft Treated Site, Autograft Comparator Site, and Normal Skin.
  Blood will be collected using EDTA, SST, PAXgene RNA and PAXgene DNA tubes for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Previous Treatment: Biologic StrataGraft Skin Tissue: This consists of areas that were treated with Stratagraft Skin Tissue under a previous clinical study STRATA2016.
  No new interventions will occur.
  Interventions: Other: Punch biopsy; Other: non-invasive photography, assessments, and measurements
- Previous Treatment: Autograft Comparator: This consists of areas that were treated with autograft comparator under a previous clinical study STRATA2016.
  No new interventions will occur.
  Interventions: Other: Punch biopsy; Other: non-invasive photography, assessments, and measurements

INTERVENTIONS:
Other: Punch biopsy — punch biopsies will be used for histologic analysis and biochemical assays
Other: non-invasive photography, assessments, and measurements — photography, scar questionnaires, pain and itch assessments, and non-invasive measurements of scar including color, stiffness, and elasticity

SUMMARY:
The purpose of this study is to describe and better understand the scars of subjects that have been treated with Stratagraft tissue vs autograft.

DETAILED DESCRIPTION:
This study will recruit patients who have previously been participants in the STRATA2016 study protocol. The patients will have comprehensive scar examinations conducted including the use of imaging, scar scale scores, pain and itch scales, scar volume measurements, and non-invasive skin measurements resulting in quantitative metrics of skin elasticity, stiffness, and color. Tissue biopsies will also be collected for histologic investigations into the scar. Each patient will have a biopsy taken of the autografted site, the Stratagraft site, and an area of normal, un-injured skin.

ELIGIBILITY:
Inclusion Criteria

1. Participant in STRATA2016 clinical trial
2. ≥ 18 years of age

Exclusion Criteria

1. Unable to provide informed consent
2. Known allergy to lidocaine
3. Scars are not appropriate for investigation based on clinical judgement by the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited using the participant enrollment records from the STRATA2016 that took place at MedStar Washington Hospital Center/MedStar Health Research Institute.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Vancouver Scar Scale scores will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
  Min value for this scale is 0 and maximum value is 13. The higher the score, the worse the scar/outcome.
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Patient and Observer Scar Assessment Scale (POSAS) scores will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
  Min value for this scale for the patient and observer components are 14 and maximum value is 140. The higher the score, the worse the scar/outcome.
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Pain visual analogue scale scores will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
  The lowest value for this scale is 0 and the highest is 100. The higher the value to worse the outcome of pain.
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Itch visual analogue scale scores will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
  The lowest value for this scale is 0 and the highest is 100. The higher the value to worse the outcome of itch.
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Non-invasive skin probe measuring color will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Non-invasive skin probe measuring elasticity will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Non-invasive skin probe measuring stiffness will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
Characterize post-burn scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Histologic measurements will be compared between scars originating from Stratagraft-treated burn wounds vs. autograft-treated burn wounds. The data will be normalized to uninjured skin.
  The specific parameters being measured include epidermal thickness (microns), dermal thickness (microns), scar cellularity (percentages), and rete ridge ratios (ratio of basement membrane length over epidermis length).

SECONDARY OUTCOMES:
Qualitatively characterize scar resulting from Stratagraft-treated and autograft-treated wounds | 1 DAY
  Digital images and 3D photography will be used to qualitatively characterize scars.
  Formalin-fixed, paraffin embedded (FFPE) samples will be used to generate sections which will be stained with Massons trichrome (overall collagen), Pircosirius red (type I and III collagen), Verhoeff Van Geison (elastin), and Fontana Masson (melanin) stains. These stained sections will be imaged and used to qualitatively characterize scar resulting from Stratagraft-treated burn wounds and SOC-treated burn wounds. Images will be normalized to uninjured skin.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States